CLINICAL TRIAL: NCT04831437
Title: Comparison of Clinical Response and Toxicity of Hypo-fractionated Chemoradiation With Standard Treatment in Patients With Uterine Cervix Cancer
Brief Title: Clinical Response and Toxicity of Hypo-fractionated Chemoradiotherapy in Cervix Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9711880002
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-03

CONDITIONS: Cervix Uteri Cancer
Keywords: Hypofractionation; Chemoradiation; Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated (Experimental): EBRT 40Gy/15fr
  Interventions: Radiation: Hypofractionated EBRT
- Control Group (Active Comparator): EBRT 45Gy/ 25fr
  Interventions: Radiation: Standard EBRT

INTERVENTIONS:
Radiation: Hypofractionated EBRT — EBRT dose of 40Gy in 15 fractions over 3 weeks plus 3 weekly infusions of cisplatin 40mg/m2
  Arms: Hypofractionated
Radiation: Standard EBRT — EBRT dose of 45Gy in 25 fractions over 5 weeks plus 5 weekly infusions of cisplatin 40mg/m2
  Arms: Control Group

SUMMARY:
Uterine cervix cancer can be treated definitively with concurrent chemoradiation (external beam radiotherapy and chemotherapy) followed by high dose rate brachytherapy. Treatment duration can be shortened by increasing the dose per fraction of treatment which can reduce costs and patient exposure. The aim of our study is to determine the non-inferiority of hypofractionated radiotherapy compared with conventional treatment.

DETAILED DESCRIPTION:
In this study we aim to determine if clinical response and toxicity of radiotherapy hypofractionation is non-inferior to the conventional treatment. We will enroll 60 eligible patients with cervical cancer stage IB to IIIC and randomly allocate them into the intervention (hypofractionation) group or the control (standard) groups. The patients in the intervention group will receive external beam radiotherapy(EBRT) to a total dose of 40 Gy in 15 fractions within 3 weeks concurrently with weekly chemotherapy with cisplatin 40mg/m2 (total of 3 cycles). Whereas, the control group will receive EBRT to a total dose of 45 Gy in 25 fractions within 5 weeks concurrently with weekly chemotherapy with cisplatin 40mg/m2 (total of 5 cycles). All patients from both groups will undergo high dose rate brachytherapy one week after completion of EBRT to a total dose of 28 Gy per 4 weekly sessions. Patients will be evaluated regarding early and late toxicities as described by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 at the completion of brachytherapy, and at 3 months, 6 months, and 3 years from completion of treatment. Also, clinical response will be evaluated through dynamic contrast enhanced pelvic MRI 3 months, 1 year, and 3 years after completion of brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathology of squamous cell carcinoma (SCC), adenocarcinoma, adenosquamous carcinoma of uterine cervix- International Federation of Gynecology and Obstetrics (FIGO) stage IB, IIA, IIB, IIIA, IIIB (due to hydronephrosis without creatinine clearance compromise), IIIC1 (if less than 3 lymph nodes with size less than 3cm, and without involvement of common iliac chain)- Patient eligible for definitive chemoradiotherapy followed by brachytherapy

Exclusion Criteria:

* Creatinine clearance less than 30ml/min, any histology other than the above, requirement of paraaortic lymph node irradiation, inflammatory bowel disease, connective tissue disorders, previous pelvic radiotherapy, FIGO stage IA or IV, Eastern Cooperative Oncology Group (ECOG) performance status greater than 2, History of previous hysterectomy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Early toxicity | 3 months after completion of treatment
  Early treatment-related toxicity within 3 months after completion of treatment as defined by CTCAE 5.0.
Early response | 3 months after completion of treatment
  Early response to treatment at 3 months after treatment completion based on dynamic contrast-enhanced pelvic MRI findings

SECONDARY OUTCOMES:
Late toxicity | 1 and 3 years after completion of treatment
  Late treatment-related toxicity within 1 and 3 years after completion of treatment as defined by CTCAE 5.0.
Progression-free survival | 5 years
  Time from randomization to progression(based on MRI and physical examination), death, or last follow up; whichever that occurs first
Disease-specific survival | 5 years
  Time from randomization to death from cervical cancer or last follow-up; whichever that occurs first.
Overall survival | 5 years
  Time from randomization to death from any reason or last follow-up; whichever that occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Maddah-Safaei, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital Complex, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maddah Safaei A, Esmati E, Gomar M, Akhavan S, Sheikh Hasani S, Malekzadeh Moghani M, Zamani N, Moshtaghi M, Malek M, Jafari F, Sharifian A, Kolahdouzan K. Hypofractionated versus standard chemoradiotherapy in the definitive treatment of uterine cervix cancer: interim results of a randomized controlled clinical trial. J Cancer Res Clin Oncol. 2024 Jan 20;150(1):20. doi: 10.1007/s00432-023-05563-8. PMID 38244105